CLINICAL TRIAL: NCT03219021
Title: Evaluation of Arch Dimensions of Children With Surgically Repaired Unilateral Cleft Lip and Palate: A Cross Sectional Study
Brief Title: Evaluation of Arch Dimensions of Children With Surgically Repaired Unilateral Cleft Lip and Palate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Menna Allah Mohammed Awad (Other)
Responsible Party: Sponsor-Investigator, Menna Allah Mohammed Awad, Master Student in department of pedodontics, Cairo University
Organization: Cairo University (Other)
Other Study IDs: CEBD-2017-7-170
Record Dates: First submitted 2017-07-09; First posted 2017-07-17 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Surgically Repaired Unilateral Cleft Lip and Palate
Keywords: Cleft lip and Palate; unilateral cleft lip and palate; surgically repaired cleft lip and palate; arch dimensions; arch discrepancies; dental arch dimensions; arch parameter; arch circumference; intercanine width; first deciduous molar width; second deciduous molar width; permanent first molar width
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess arch dimensions among children with surgically repaired unilateral cleft lip and palate.

DETAILED DESCRIPTION:
Measurements of arch widths will be performed in the maxillary and mandibular arches after performing a study cast. Alginate impression of the upper and lower arch of all participating children will be performed and poured immediately to prevent dimensional changes.

The inter-deciduous canine, inter-permanent molar, and the distances between the first and second deciduous molars will be measured using a digital caliper directly on dental casts by a single examiner.

Distance measurements will be obtained between cusp tips of canines, cusp tips of first deciduous molars, mesiobuccal cusp tips of second deciduous molars, and mesiobuccal cusp tips of first permanent molars. Estimated cusp tips will be used in cases of wear facets.

Rationale:

Children with cleft lip and/or palate suffer from problems in growth of the jaws, particularly the maxilla (upper jaw), as a result of surgical repairs of the cleft lip and palate. It is important to know the arch dimensions of them to enable the identification of specific surgical alterations related to maxillofacial growth concerning the common treatment protocol for patients with cleft lip and palate.

Benefits to the practitioner:

-Increase the awareness of pediatric dentists about changes of arch dimensions of surgically repaired cleft lip and palate patients in Egypt.

Benefits to the patient:

* Inform parents about any disturbances that might be associated with Cleft lip and Palate.
* Guide them to the orthodontic care if needed.

Benefits to the community:

* Provide the Egyptian community with data concerning patients with cleft lip and palate.
* Increase awareness of problems related to Cleft Lip and Palate.

ELIGIBILITY:
Inclusion Criteria:

* Children with cleft lip and palate from the age group: 8-10 years.
* Unilateral Cleft lip and palate children.
* Children who had been operated with lip and palate closure

Exclusion Criteria:

* Cleft lip and palate patients with systemic diseases, autoimmune conditions, syndromes.
* Children with any arch expansion or orthodontic procedure or previous history of orthodontic treatment.
* The presence of early loss of deciduous molars.
* Parents refusing participation in the study

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with surgically repaired unilateral cleft lip and palate
Sampling Method: Non-Probability Sample
Enrollment: 233 (Estimated)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
arch dimensions measures | Day 1
  Assessment of arch dimensions among children with surgically repaired unilateral cleft lip and palate in mm using digital caliper